CLINICAL TRIAL: NCT03297749
Title: Genetic Variants and Oxidative Stress as Links Between Periodontitis and Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: University of Catania (Other)
Responsible Party: Sponsor
Other Study IDs: 4242/01
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Periodontitis, Adult; Metabolic Syndrome
MeSH Terms: conditions — Chronic Periodontitis; Metabolic Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study (no intervention) — No interventions
  Other Names: No interventions

SUMMARY:
The aim of this study is to investigate the systemic impact of periodontitis in patients with Metabolic Syndrome, by assessing measures of sub-clinical atherosclerosis and cardiovascular risk, microbial factors and host genetic variants, and to study the possible effect of mediators of inflammation and oxidative stress as links between the two conditions.

DETAILED DESCRIPTION:
This is a cross-sectional study. 102 patients with metabolic syndrome will be recruited and will have periodontal and dental examination for diagnosis of caries and periodontal diseases. They will undergo blood, saliva, GCF and subgingival plaque sampling and a series of tests on cardiovascular disease, including measures of pulse-wave velocity,carotid intima-media thickness and echocardiography assessment. Statistical analysis will assess associations between dental diagnoses and metabolic, cardiovascular, inflammatory, genetic, microbial and cardiovascular risk outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* Age 18- 75
* Diagnosis of metabolic syndrome
* Presence of at least 12 teeth

Exclusion Criteria:

* Pregnancy
* Presence of infectious diseases such as hepatitis and HIV
* Use of non-steroidal anti-inflammatory drugs (excluding low-dose aspirin) within one month prior to the baseline visit
* Use of systemic antibiotics within three months prior to the baseline visit
* Antibiotic pre-medication required for the performance of periodontal examination

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with metabolic syndrome will be recruited from outpatients attending the Internal Medicine Unity at the University of Catania.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
pulse wave velocity | baseline
oxidative stress | baseline
carotid intima-media thickness | baseline
genetic variants | baseline
left ventricular mass | baseline

SECONDARY OUTCOMES:
inflammatory markers | baseline
subgingival microbes | baseline

CONTACTS AND LOCATIONS:
Locations (2):
- University of Catania, Catania, Italy
- UCL, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nibali L, Donos N, Terranova V, Di Pino A, Di Marca S, Ferrara V, Pisano M, Scicali R, Rabuazzo AM, Purrello F, Malatino L. Left ventricular geometry and periodontitis in patients with the metabolic syndrome. Clin Oral Investig. 2019 Jun;23(6):2695-2703. doi: 10.1007/s00784-018-2667-8. Epub 2018 Oct 22. PMID 30350134